CLINICAL TRIAL: NCT02401412
Title: A Study Determining Variances in Ostomy Skin Conditions And The Economic Impact.
Brief Title: The Advocate Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hollister Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 5787-O
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Ostomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Ostomy Barrier (Other): The test product is a new Hollister ostomy barrier.
  Interventions: Device: Test Ostomy Barrier
- Control Ostomy Barrier (Other): The control product is a currently marketed Hollister ostomy barrier.
  Interventions: Device: Control Ostomy Barrier

INTERVENTIONS:
Device: Test Ostomy Barrier
  Arms: Test Ostomy Barrier
Device: Control Ostomy Barrier
  Arms: Control Ostomy Barrier

SUMMARY:
Hollister Incorporated is studying stoma related cost of care related to a new ostomy skin barrier that is designed to maintain adhesive properties and good peristomal skin health compared to other currently marketed barriers.

ELIGIBILITY:
Inclusion Criteria:

Ostomy patients who:

* Have healthy peristomal skin
* Are within 12 weeks post op

Exclusion Criteria:

Ostomy patients who:

* Have a fistula, wound, lesion or suspected infection in the peristomal area
* Are in-patient in healthcare facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kalifa, Study Director — Hollister Incorporated
Locations (12):
- United States (8):
  - Stoia Consultants, Riverside, California
  - Jupiter Medical Center, Jupiter, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - Indiana Health Ball Memorial University, Muncie, Indiana
  - Restored Images, Kansas City, Missouri
  - Klein's Orthopedic & Medical Supply, Cuyahoga Falls, Ohio
  - St. Elizabeth Hospital, Youngstown, Ohio
- Canada (4):
  - Lakeside Medicine Center, Kelowna, British Columbia
  - Pharmasave, Nanaimo, British Columbia
  - Ostomy Care Centre, New Westminster, British Columbia
  - Rouge Valley Health System, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Ostomy Barrier: The test product is a new Hollister ostomy barrier.
  Test Ostomy Barrier
- Control Ostomy Barrier: The control product is a currently marketed Hollister ostomy barrier.
  Control Ostomy Barrier
Period: Overall Study
Arm/Group | Test Ostomy Barrier | Control Ostomy Barrier
Started | 89 | 81
Received Study Device | 89 | 80
Completed | 59 | 49
Not Completed | 30 | 32
Not completed — Lost to Follow-up | 1 | 0
Not completed — Discontinued Intervention | 15 | 21
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Subject withdrawal prior to intervention | 0 | 1
Not completed — Improper Enrollment per In/Ex Criteria | 10 | 6

BASELINE CHARACTERISTICS:
Population: The analysis population was defined as a modified ITT population which excluded subjects who
  1. were inappropriately enrolled into the study (i.e. subjects initially enrolled but later found to NOT meet inclusion/exclusion criteria); (n=16)
  2. did not receive the study device; (n=1)
  As such 153 (170-17) subjects were eligible for analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Ostomy Barrier | Control Ostomy Barrier | Total
Number analyzed (Participants) | 79 | 74 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (24.8) | 57.2 (15.2) | 56.3 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 60
  Male | 50 | 43 | 93
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 15 | 12 | 27
  United States | 56 | 53 | 109
  Europe | 8 | 9 | 17
BMI [Mean (Standard Deviation); unit: kg/m2] | 24.8 (5.8) | 26.4 (5.8) | 25.6 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Stoma Related Cost of Care
Description: 12 week stoma related cost of care. Cost of care includes treatments related to ostomy and/or PSCs (topical medications, clinic visits, and selected accessory use), social impact of ostomy and/or PSCs (missed work/ appointments), ostomy-related hospitalizations, emergency department visits, physician/clinic visits, medication use and therapies, and product utilization.
Time Frame: 12 weeks
Population: as for baseline characteristics
Measure: Least Squares Mean (95% Confidence Interval); unit: USD
Arm/Group | Test Ostomy Barrier | Control Ostomy Barrier
Number analyzed (Participants) | 79 | 74
USD | 223.73 [210.86 to 236.60] | 260.19 [242.79 to 277.58]

2. Secondary Outcome: Peristomal Skin Complication Rate
Description: Observed 8 week Peristomal Skin Complication (PSC) rate. The validated Ostomy Skin Tool DET score was used to describe the status of the peristomal skin. Subjects were deemed to have had a PSC if the DET score was above zero due to anything other than normal postoperative healing and/or scar tissue, or the DET score increased above the normal score obtained at a previous visit.
Time Frame: 8 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Test Ostomy Barrier | Control Ostomy Barrier
Number analyzed (Participants) | 79 | 74
Participants | 32 | 41

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse Events were determined via standardized study investigator assessment forms. All Adverse Events are reported irrespective of relation to study product.
  Adverse Events were reported for the modified ITT population which excluded subjects who
  1. were inappropriately enrolled into the study (i.e. subjects initially enrolled but later found to NOT meet inclusion/exclusion criteria); (n=16)
  2. did not receive the study device; (n=1)
  As such AEs reported for 153 (170-17) subjects
Arm/Group | Test Ostomy Barrier | Control Ostomy Barrier
All-Cause Mortality (participants affected / at risk) | 2/79 | 0/74
Serious Adverse Events (participants affected / at risk) | 12/79 | 6/74
Other Adverse Events (participants affected / at risk) | 6/79 | 11/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Ostomy Barrier (N=79) | Control Ostomy Barrier (N=74)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0
Death due to septic shock (Infections and infestations) | 1 (1) | 0
Pelvic Abscess (Infections and infestations) | 1 (1) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0
Intestinal Blockage/Illeus (Gastrointestinal disorders) | 4 (4) | 1 (1)
Acute shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0
Death due to primary cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0
Inflamed gall bladder (Gastrointestinal disorders) | 0 | 1 (1)
Non-specific Failure to Thrive (General disorders) | 0 | 1 (1)
Non-specific Pain (Renal and urinary disorders) | 0 | 1 (1)
Cellulitis (Infections and infestations) | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Ostomy Barrier (N=79) | Control Ostomy Barrier (N=74)
Elective colonoscopy (Surgical and medical procedures) | 1 (1) | 0
Incisional Abscess (Infections and infestations) | 1 (1) | 0
Intestinal Blockage/Illeus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stoma abrasion caused by patient (Injury, poisoning and procedural complications) | 1 (1) | 0
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Ostomy pouching system not secure (Product Issues) | 1 (1) | 0
Peristomal Skin Complication (Skin and subcutaneous tissue disorders) | 0 | 7 (7)
Stoma complication (Gastrointestinal disorders) | 0 | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT02401412/Prot_SAP_000.pdf